CLINICAL TRIAL: NCT04788407
Title: Pilot Study of Safety and Efficacy of Nitazoxanide in Post-exposure Prophylaxis in Household Contacts of Patients With Confirmed SARS-CoV-2 Infection
Brief Title: Efficacy and Safety of Nitazoxanide for Post Exposure Prophylaxis of COVID-19 in Household Contacts
Acronym: PENTZ
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Huésped (Other)
Collaborators: Ministerio de Salud de Ciudad Autónoma de Buenos Aires (Other Government); Laboratorios Roemmers S.A.I.C.F. (Industry)
Responsible Party: Principal Investigator, Omar Sued, Research Director, Fundación Huésped
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FH-53
Record Dates: First submitted 2021-03-07; First posted 2021-03-09 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Covid19; SARS-CoV-2 Infection; Households Contacts
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Prospective, Cluster-Randomized, double-blind, placebo-controlled clinical trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Experimental): Subjects will receive nitazoxanide 500 mg TID.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Subjects will receive placebo TID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Subjects will receive nitazoxanide 500 mg TID for 7 days
  Other Names: Nixoran
  Arms: Nitazoxanide
Drug: Placebo — Subjects will receive placebo TID for 7 days
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the drug nitazoxanide 500 mg, administered three times a day, in relation to placebo in preventing the development of COVID-19 in household contacts of patients diagnosed with the disease.

DETAILED DESCRIPTION:
Eligible participants (cohabitants of a recently confirmed COVID19 case) residing in Buenos Aires City will be identified by the Ministry of Health and contacted with the investigators, who will visit them at home and offer to participate. For consenting individuals, a rapid serological test and a nasopharyngeal PCR sample for SARS-CoV-2 will be performed and participants will be then randomized to NTZ or placebo to be taken during 7 days.

SARS-CoV-2 PCR will be repeated on day 14th and the serologic rapid test repeated on day 28th.

Clinical status of participants will be assessed daily by phone. Individuals meeting case definition will be evaluated at home and a PCR will be performed. Those with confirmed COVID19 case will discontinue study medication and followed until symptoms resolution.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 and under 65.
* Household contact with a confirmed case of COVID-19 by PCR for Sars-CoV-2.
* Initiate study medication within 4 days from the last close contact with the index case.
* The patient must not present symptoms suggestive of Covid19 (cough, dyspnea, fever> 37.5 C, fatigue, sore throat, myalgia, diarrhoea) at the time of admission to the study and from previous 14 days.
* Informed consent from the patient or legal representative.

Exclusion Criteria:

* History of infection confirmed by SARS-CoV-2.
* Positive IgG antibodies test for SARS-CoV-2 at the time of admission.
* Have received any dose of nitazoxanide within 7 days prior to screening.
* Known hypersensitivity to any of the study medication components.
* Use of any investigational or unregistered drug or vaccine within 30 days prior to screening, or use planned during the study period.
* Inability to comply with study procedures.
* Current breastfeeding.
* Pregnancy.
* Intolerance or inability to take oral medication.
* History of severe liver disease (Child-Pugh B or C) and/or chronic kidney disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with laboratory-confirmed COVID-19 identified after start of treatment and before the end of the study | 28 days
  Proportion of participants with negative baseline PCR for SARS-CoV-2 who test positive for PCR on day 14 and / or seroconversion on day 28 after initiation of study medication.

SECONDARY OUTCOMES:
Proportion of adverse events (AE) and serious AE (SAE) related to research product. | 28 days
  Safety and adverse events (AEs).
Incidence of all causes of study drug withdrawal or discontinuation. | 7 days
  Treatment adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Sued, MD PhMD, Study Director — Fundacion Huesped.; Herman K Ludvik, MD, Principal Investigator — Fundación Huésped
Locations (1):
- Fundación Huésped., Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes
to publish study results
URL: https://www.huesped.org.ar/que-hacemos/ciencia/investigaciones-biomedicas/